CLINICAL TRIAL: NCT01819246
Title: High Yield Intraoperative, Autologous Platelet Apheresis-Optomizing Transfusion Practice In Cardiac Surgery
Brief Title: High Yield Intraoperative, Autologous Platelet Apheresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00011798
Record Dates: First submitted 2013-02-19; First posted 2013-03-27 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Allogenic Transfusion of Platelets During Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pheresis Treatment Arm (Active Comparator)
  Interventions: Procedure: Aphersis Treatment Arm
- Control Arm (Sham Comparator)
  Interventions: Other: Control Arm

INTERVENTIONS:
Procedure: Aphersis Treatment Arm
  Arms: Pheresis Treatment Arm
Other: Control Arm
  Arms: Control Arm

SUMMARY:
The overall aim is to reduce overall allogeneic transfusion requirements during cardiac surgery when compared to standard management.

To evaluate this the investigators will test the hypothesis that intraoperative, autologous platelet apheresis will primarily avoid allogeneic platelet transfusion. Following induction of anesthesia and intravascular line insertion, the patient will be randomized to control or treatment arms by sealed envelope technique where computer generated, randomization numbers are assigned prior to enrollment based on study patient number which is never reused.

The control arm will have central venous access "sham" connected to the apheresis machine Trima® (Terumo BCT, Denver CO); the treatment arm will be connected and undergo pheresis. The clinical team will be blinded by a sterile sheet acting as a curtain and a recorded playback of the typical sounds of the operation of the apheresis machine. At the end of the pheresis, the platelet units will be disguised with opaque coverings and agitated at room temperature in compliance with the American Association of Blood Banks (AABB) recommendations for platelet storage. On separation from CPB, the blinded administration of autologous platelets or allogeneic (blood bank) platelets will occur after protamine administration, if the surgeon requests platelet transfusion (this is typically the case for these operations). The surgeon will be blinded and he will order subsequent transfusions based on clinical evidence of microvascular bleeding in accordance with standard guidelines, as is the investigators practice for these operations.

ELIGIBILITY:
Inclusion Criteria:

* All elective, aortic reconstruction surgery and other patients at high risk of receiving platelet transfusions such as: combined CABG/valve, more than one valve surgery via median sternotomy, left ventricular assist devise, and pulmonary thromboarterectomy with deep hypothermic circulatory arrest cases.
* Over 18 years of age

Exclusion Criteria:

* renal disease (dialysis dependent, end-stage renal disease or a baseline Cr >3mg/dl)
* known coagulopathy/bleeding tendency (such as von Willebrand disease)
* platelet count of <150x109 /liter at baseline
* Hct < 30%
* platelet inhibitory drugs within 5 days prior to surgery or Aspirin 325 mg within 48 hrs of surgery
* inability to provide written, informed consent
* patients receiving pre-operative parenteral, non-heparin anticoagulants will be excluded
* pregnancy is not an exclusion criterion for the study but, typically, pregnancy is a contraindication to elective cardiac surgery hence pregnant patients are unlikely to be encountered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of allogeneic platelet units transfused. | During the operative procedure

SECONDARY OUTCOMES:
Overall blood product transfusion. | During the operative procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ian Welsby, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Mathew JP, Grocott HP, Phillips-Bute B, Stafford-Smith M, Laskowitz DT, Rossignol D, Blumenthal JA, Newman MF; Neurologic Outcome Research Group of the Duke Heart Center; Cardiothoracic Anesthesiology Research Endeavors Investigators of the Duke Heart Center. Lower endotoxin immunity predicts increased cognitive dysfunction in elderly patients after cardiac surgery. Stroke. 2003 Feb;34(2):508-13. doi: 10.1161/01.str.0000053844.09493.58. PMID 12574568
- [Background] Ford SM, Unsworth-White MJ, Aziz T, Tooze JA, van Besouw JP, Bevan DH, Treasure T. Platelet pheresis is not a useful adjunct to blood-sparing strategies in cardiac surgery. J Cardiothorac Vasc Anesth. 2002 Jun;16(3):321-9. doi: 10.1053/jcan.2002.124141. PMID 12073204